CLINICAL TRIAL: NCT02685956
Title: Clinical Evaluation of the Sentosa SA HSV1/2 Qualitative PCR Test
Status: Completed | Type: Observational
Sponsor: Vela Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: Vela Sentosa HSV Study
Record Dates: First submitted 2016-02-10; First posted 2016-02-19 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Herpes Simplex
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples collected from an oral or genital site, submitted to a clinical laboratory for the purpose of testing for the presence of HSV1 or HSV2.
  Samples collected in universal viral transport media, using a plastic shaft swab made of either polyester, cotton, rayon or Dacron.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vela Sentosa SA HSV1/2 PCR Test: Male and female subjects of any age with sample collected from a lesion and submitted to a clinical laboratory for the purpose of testing for the presence of HSV1 or HSV2 and diagnosing HSV infection.
  Interventions: Device: Vela Sentosa SA HSV1/2 Qualitative PCR Test

INTERVENTIONS:
Device: Vela Sentosa SA HSV1/2 Qualitative PCR Test — medical device test using Vela Sentosa SA HSV1/2 Qualitative PCR Test
  Other Names: Sentosa HSV Assay

SUMMARY:
The purpose of this study is to evaluate the performance of the Sentosa SA HSV1/2 Qualitative PCR Test. Precision of results and concordance of results with a reference assay will be evaluated.

DETAILED DESCRIPTION:
This study will utilize residual samples from male and female patients with signs and symptoms of oral or genital HSV infections. Genital samples will include internal and external genital lesions such as those collected from lesions of the anus, buttocks, vagina, labia, or penis. Oral samples will include those collected from lip, gum, and mouth lesions. For concordance testing, the sample size is based on historical study design and estimates of the expected prevalence of HSV1 and/or HSV2 in the population enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Sample was taken from a lesion from an internal or external oral or genital site.
* Sample was submitted to a clinical laboratory for the purpose of testing for the presence of HSV1 or HSV2.
* The following information about the patient from which the sample was taken is available: presumptive diagnosis or signs and symptoms causing assay requisition; site of lesion; age at time of sample collection or date of birth, and sex.
* Sample was collected in universal viral transport media, using a plastic shaft swab made of either polyester, cotton, rayon or Dacron.
* There is sufficient residual sample to perform both test and reference assays.

Exclusion Criteria:

* Sample leaked during shipment or storage prior to assay.
* Sample has undergone more than 1 freeze-thaw cycle before testing;
* Sample eluent is not clear after centrifugation (refer to section 6.3.1).
* Sample ID is missing or ambiguous.
* Sample is collected using alginate calcium swab.
* Sample handling and storage requirement in section 5.4 not followed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and females with genital or oral lesions to be tested for HSV 1/2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 2295 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaw Chiat Hong, Study Director — Vela Diagnostics
Locations (9):
- United States (9):
  - Tampa General Hospital, Tampa, Florida
  - Baystate Health, Springfield, Massachusetts
  - Beaumont Health, Royal Oak, Michigan
  - BioReference Labs, Elmwood Park, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Geisinger Health, Danville, Pennsylvania
  - Quest Diagnostics, Horsham, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - MedFusion, Lewisville, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vela Diagnostics Website — http://www.veladx.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Lesions: Male and female subjects of any age with sample collected from an oral lesion and submitted to a clinical laboratory for the purpose of testing for the presence of HSV1 or HSV2 and diagnosing HSV infection.
- Anogenital Lesions: Male and female subjects of any age with sample collected from an anogenital lesion and submitted to a clinical laboratory for the purpose of testing for the presence of HSV1 or HSV2 and diagnosing HSV infection.
Period: Overall Study
Arm/Group | Oral Lesions | Anogenital Lesions
Started | 317 | 1978
Completed | 317 | 1978
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Lesions | Anogenital Lesions | Total
Number analyzed (Participants) | 317 | 1978 | 2295
Age, Customized [Count of Participants; unit: Participants]
  0 - 10 | 54 | 64 | 118
  11 - 20 | 31 | 275 | 306
  21 - 30 | 66 | 684 | 750
  31 - 40 | 40 | 378 | 418
  41 - 50 | 25 | 257 | 282
  51 - 60 | 34 | 170 | 204
  61 - 70 | 32 | 91 | 123
  71 - 80 | 28 | 41 | 69
  81 - 90 | 7 | 15 | 22
  >90 | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 1573 | 1753
  Male | 137 | 405 | 542
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 317 | 1978 | 2295

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Positive and Negative for HSV-1 by SA201 HSV-1/2 PCR Test
Description: Study will assesses Sentosa HSV 1/2 assay fpr detecting HSV DNA compared to traditional microbiology culture-based ELVIS method (reference assay). HSV DNA detection is determined for each virus (HSV 1 and 2) at each type of anatomic site (genital lesion and oral lesion).
Time Frame: within 60 days of last sample enrollment
Population: Analysis group included samples from 290 anogenital and 1291 anogenital lesions tested for HSV1 using the ELVIS HSV ID and D3 Typing Test System (N=1581). A further 397 that tested HSV2 positive by ELVIS were excluded from the HSV1 analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Anogenital Lesions With POSITIVE HSV1 ELVIS Result: Sample collected from an anogenital lesion and tested positive for HSV1 using the ELVIS HSV ID and D3 Typing Test System (ELVIS)
- Anogenital Lesions With Negative HSV1 ELVIS Result: Sample collected from an anogenital lesion and tested negative for HSV1 using the ELVIS HSV ID and D3 Typing Test System (ELVIS)
Arm/Group | Anogenital Lesions With POSITIVE HSV1 ELVIS Result | Anogenital Lesions With Negative HSV1 ELVIS Result
Number analyzed (Participants) | 290 | 1291
Participants
  HSV-1 POSITIVE by SA201 HSV-1/2 PCR Test | 281 | 54
  HSV-1 NEGATIVE by SA201 HSV-1/2 PCR Test | 9 | 1237

2. Primary Outcome: Number of Participants Positive and Negative for HSV-2 by SA201 HSV-1/2 PCR Test
Description: Study asses Sentosa HSV 1/2 assay in detecting HSV DNA compared to traditional microbiology culture-based ELVIS method (reference assay). HSV DNA detection is determined for each virus (HSV 1 and 2) at each type of anatomic site (genital lesion and oral lesion).
Time Frame: within 60 days of last sample enrollment
Population: Analysis group included samples from N=1978 anogenital lesions tested for HSV2 using the ELVIS HSV ID and D3 Typing Test System.
Measure: Count of Participants; unit: Participants
Groups:
- Anogenital Lesions With POSITIVE HSV2 ELVIS Result: Sample collected from an anogenital lesion and tested positive for HSV2 using the ELVIS HSV ID and D3 Typing Test System (ELVIS)
- Anogenital Lesions With NEGATIVE HSV2 ELVIS Result: Sample collected from an anogenital lesion and tested negative for HSV2 using the ELVIS HSV ID and D3 Typing Test System (ELVIS)
Arm/Group | Anogenital Lesions With POSITIVE HSV2 ELVIS Result | Anogenital Lesions With NEGATIVE HSV2 ELVIS Result
Number analyzed (Participants) | 397 | 1581
Participants
  HSV-2 POSITIVE by SA201 HSV-1/2 PCR Test | 391 | 147
  HSV-2 NEGATIVE by SA201 HSV-1/2 PCR Test | 6 | 1434

ADVERSE EVENTS:
Time Frame: This trial utilized remnant laboratory specimens and all results were monitored for accuracy and adverse events upon the completion of the testing phase of the study.
Description: This is a remnant sample study using leftover HSV swab sample media. All case data was fully monitored on completion of the testing phase of the study and no adverse events associated with study subjects contributing biospecimens were identified..
  There was also reporting mechanism in place to record device user adverse events however no in vitro diagnostic device user adverse events were reported in the study
Arm/Group | Oral Lesions | Anogenital Lesions
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has 45 days to review and comment. Sponsor may extend the embargo period for no more than an additional 60 days in order to file a patent application due to patentable subject matter contained in the proposed presentation or publication. If the Sponsor objects to the publication or presentation due to the existence of confidential information, the institution shall remove the confidential information before disclosure.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT02685956/Prot_SAP_000.pdf